CLINICAL TRIAL: NCT03108404
Title: Predictive Score for Neonatal Mortality for Women With Premature Rupture of Membranes Between 22 and 28 Weeks of Gestation
Acronym: PPROM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2016-13 Pr Tourneux-3
Record Dates: First submitted 2017-03-31; First posted 2017-04-11 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Perinatal Mortality; Premature Rupture of Fetal Membranes
Keywords: predictive score
MeSH Terms: conditions — Perinatal Death; Fetal Membranes, Premature Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Validation of a diagnostic test — Validation of a diagnostic test

SUMMARY:
Pretern premature rupture of the membranes (PPROM) remains the leading cause of preterm deliveries and neonatal mortality and morbidity. PPROM is defined as rupture of the fetal membranes prior to 37 weeks' gestation. PPROM complicates 2-4% of all pregnancies and accounts for approximately 30 % of preterm births.

The etiology of PPROM remains elusive. PPROM is one of the main causes of prematurity and its complications, such as newborn respiratory distress syndrome, neonatal sepsis, necrotizing enterocolitis, intraventricular hemorrhage, perventricular leucomalacia, varying degrees of lung hypoplasia and bronchopulmonary dysplasia. All these factors contribute greatly to an increase in neonatal morbidity and mortality Management of PPROM followed actual guidelines. Conservative management to prolong a pregnancy is a classical approach to treat PPROM before 34 weeks' gestation in association with antibiotic therapy and corticosteroids.

Maternal and neonatal data were collected from maternal and newborns medical records.

ELIGIBILITY:
Inclusion Criteria:

* Women with PPROM between 22 weeks and 27 weeks and 6 days are eligible for this study

Exclusion Criteria:

* Therapeutic abortion / terminaison of pregnancy
* Intra uterine demise
* active labor with cervical dilatation of 3 cm with regular contractions.
* Triplet pregnancies

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with premature rupture of membranes between 22 + 0 and 27 + 6 SA included
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-06 (Estimated); Study Completion 2020-01-06 (Estimated)

PRIMARY OUTCOMES:
The purpose was to determine which antepartum criteria were efficient to predict neonatal death, in order to create a predictive prognostic antenatal index of mortality. | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France